CLINICAL TRIAL: NCT03606434
Title: Sex Differences in Reflex Responses to Intermittent Hypoxia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Missouri-Columbia (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Jacqueline K Limberg, PhD, Assistant Professor, University of Missouri-Columbia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2011312; 4R00HL130339 (NIH)
Record Dates: First submitted 2018-06-11; First posted 2018-07-30 (Actual); Last update posted 2021-07-21 (Actual); Status verified 2021-07

CONDITIONS: Healthy Participants

STUDY DESIGN:
Intervention Model Description: All participants will undergo same 30 minute intermittent hypoxia protocol.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Hypoxic Exposure (Experimental): Men, and women in early or late follicular phase of menstrual cycle will be exposed to acute and intermittent hypoxic episodes.
  Interventions: Other: Hypoxic exposure

INTERVENTIONS:
Other: Hypoxic exposure — 30 minutes of intermittent hypoxia

SUMMARY:
The purpose of the present study is to determine whether there are sex differences in the reflex responses to hypoxia in humans.

DETAILED DESCRIPTION:
Over 35% of the US population will develop sleep apnea at some point in their life. Sleep apnea is the most common form of sleep disordered breathing and patients with sleep apnea are at increased risk of developing high blood pressure. Intermittent, repeated exposures to low oxygen during sleep (intermittent hypoxia, IH) has been implicated as the primary stimulus for increases in sympathetic nervous system activity and blood pressure with sleep apnea. Interestingly there are some reports of a lower incidence of hypertension in women with sleep apnea when compared to men. Results from the present study will provide information important to the investigator's understanding of potential sex-differences in clinical outcomes for conditions related to acute/chronic hypoxia and may have important implications for treatments which may improve blood pressure control in patients with sleep apnea.

ELIGIBILITY:
Inclusion Criteria:

* healthy adult men and women;
* BMI <30 kg/m2;
* non-pregnant;
* non-breastfeeding;
* non-smokers;
* premenopausal women with a normal menstrual cycle unaffected by hormonal contraceptive use;
* taking no medications known to affect autonomic or cardiovascular function (PI discretion).

Exclusion Criteria:

* taking any medications known to affect the cardiovascular or autonomic nervous system (e.g. alpha-blockers, beta-blockers, etc);
* a self-reported history of hepatic, renal, pulmonary, cardiovascular, or neurological diseases;
* stroke or neurovascular disease;
* bleeding/clotting disorder;
* sleep apnea or other sleep disorders;
* diabetes;
* smoking;
* history of alcoholism or substance abuse;
* hypertension.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2018-09-13 (Actual); Primary Completion 2021-07-15 (Actual); Study Completion 2021-07-15 (Actual)

PRIMARY OUTCOMES:
Change from baseline Hypoxic Ventilatory Response after intermittent hypoxia | Through completion of intermittent hypoxia, an average of 3 hours
  Hypoxia breathing will be recorded before and after intermittent hypoxia
Change from baseline Blood Pressure after intermittent hypoxia | Through completion of intermittent hypoxia, an average of 3 hours
  Systolic and diastolic blood pressure will be recorded before and after intermittent hypoxia
Change from baseline Forearm Blood Flow after intermittent hypoxia | Through completion of intermittent hypoxia, an average of 3 hours
  Blood flow in the forearm will be recorded before and after intermittent hypoxia

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Limberg, PhD, Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri-Columbia, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No